CLINICAL TRIAL: NCT00427778
Title: The Treatment of Stress Urinary Incontinence Using an Incontinence Ring: A Randomized, Cross-over Trial
Brief Title: Incontinence Ring on Stress Urinary Incontinence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Queen's University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Dr. Marie-Andree Harvey, Principal Investigator, Queen's University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: obgy-160-06
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Stress Urinary Incontinence; Urinary Incontinence
Keywords: incontinence ring; pessary; urinary incontinence; urodynamic study; quality of life; crossover trial; randomised trial
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Incontinence ring then no intervention (Experimental): Participants first were fitted with an incontinence ring, which they wore continuously for 4 weeks. The ring wa then removed and a washout period of 2 weeks followed. Then the second 4-week period with no ring was completed.
  Interventions: Device: incontinence ring
- No intervention then incontinence ring (Experimental): Participants spend the first study 4-week period with no intervention. Then, a wasout period of 2 weeks followed. Participants were then fitted with an incontinence ring, which they wore continuously for 4 weeks.
  Interventions: Device: incontinence ring

INTERVENTIONS:
Device: incontinence ring — Incontinence ring fitted to patient's anatomy (by choosing appropriate size). It is worn continually for the duration of the treatment period.
  Intravaginal incontinence ring placed proximally in the posterior vaginal fornix. Knob located at mid-urethra.
  Other Names: Silicone Flexible Pessary; Milex code: KPCON

SUMMARY:
This study aims as defining success rate of the incontinence ring in women with test proven stress urinary incontinence and determining factors associated with successful use.

DETAILED DESCRIPTION:
The primary objective of this study is to determine if the incontinence ring is effective in decreasing the incontinence episode frequency per week. Other objectives include the determination of the cure rate (objective and subjective) with the ring, the effects to bladder function as noted on urodynamic testing, the impact on quality of life and the acceptability to this device in the treatment of stress urinary incontinence.

In this cross-over study, 40 women will undergo a two-period treatment. In one of the periods, she will spend 4 weeks wearing continuously the ring and in the other (also 4 weeks duration), she will not be using any treatment for her incontinence. Between periods, she will spend 2 weeks in "wash out" to eliminate the risk of continuous effect from the treatment in the preceding period. Each woman will be randomly assigned to the treatment sequence.

Stress urinary incontinence is a common problem affecting at almost 20% of women. Treatments currently advocated include pelvic floor exercises and surgery. Pelvic floor exercises require great motivation and usually 3 months of training to show an impact. Surgery is very effective, but costly and carries a number of complications. The use of the incontinence ring may allow women to control their symptoms with immediate result at minimal risk. This device has never been properly evaluated before its introduction into the market.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of urinary stress urinary incontinence (i.e. urinary leakage associated with increased intra-abdominal pressure/cough) (if mixed incontinence the urinary stress urinary incontinence symptoms must predominate)
* Urodynamic Stress urinary incontinence confirmed by urodynamic studies (i.e. urinary leakage associated with increased intra-abdominal pressure/cough in the absence of detrusor overactivity)
* Ability to understand spoken and written English

Exclusion Criteria:

* Severe pelvic organ prolapse (> or = stage 3 on the Pelvic Organ Prolapse Quantification System - POP-Q)
* Contraindications to pessary use (including acute vaginal/urinary or pelvic infections, vaginal or cervical lesions or unexplained vaginal bleeding)
* Inability to properly fit the incontinence ring

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Andree Harvey, MD MSc, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 87 women were screened for eligibility between June 2006 and February 2008, at an academic specialty center
Pre-assignment Details: 29 out of 87 were randomised. of those not randomized, 52 declined to participate and 6 did not meet inclusion criteria.
Groups:
- Incontinence Ring, Then no Treatment: participants first were fitted to an incontinence ring, which they wore for a period of 4 weeks, then it was removed. After a washout period of 2 weeks, they continued evaluation but with no active treatment
- No Treatment, Then Incontinence Ring: Participants first were assessment while no active treatment was received, for a period of 4 weeks. After a washout period of 2 weeks, they continued evaluation after an incontinence ring was fitted.
Period: First Intervention (4 Weeks)
Arm/Group | Incontinence Ring, Then no Treatment | No Treatment, Then Incontinence Ring
Started | 14 | 15
Completed | 10 | 14
Not Completed | 4 | 1
Not completed — no longer interested | 1 | 0
Not completed — Not successfully fitted with ring | 2 | 0
Not completed — unable to manipulate ring due to OA | 0 | 1
Not completed — anxious about using ring | 1 | 0
Period: Wash Out (2 Weeks)
Arm/Group | Incontinence Ring, Then no Treatment | No Treatment, Then Incontinence Ring
Started | 10 | 14
Completed | 10 | 14
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Incontinence Ring, Then no Treatment | No Treatment, Then Incontinence Ring
Started | 10 | 14
Completed | 10 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: all patients who were recruited and for whom a pessary was fitted, successfully or not.
Groups:
- All Study Participants: All participants who were randomised to a treatment sequence group
Arm/Group | All Study Participants
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29 (6.8)
Parity [Median (Inter-Quartile Range); unit: previous vaginal births] — number of previous vaginal birth
  previous vaginal births | 2 [1.5 to 3]
Smoking status [Count of Participants; unit: Participants] — Current smokers
  Participants | 2
Menopausal status [Count of Participants; unit: Participants] — number of women who are postmenopausal at time of study entry
  Participants | 8
Pop stage [Count of Participants; unit: Participants] — number of women at each POPQ stage. The pelvic organ prolapse quantification system is a validated method to measure prolapse in each vaginal compartments (ant, post and apical). It assesses the distance of predetermined vaginal points from the hymen during valsalva. It is divided in 5 stages: 0 (no support defect, apex no more than 'total vaginal length' minus 2 cm from hymen), 1 (leading edge >1cm above the hymen), 2 (within one cm inside or outside the hymen), 3 (more than one cm below hymen, 4 (completely out, apex more than 'total vaginal length' minus 2 cm outside from hymen)
  Participants
    stage 0 | 2
    stage 1 | 7
    stage 2 | 17
incontinence episodes per week [Median (Inter-Quartile Range); unit: number of incontinence episodes per week] | 10 [5 to 28]
Score to question #3 on UDI-6 [Median (Inter-Quartile Range); unit: units on a scale] — Score (0-3) of response to question #3 (stress incontinence specific) of Urogenital Distress inventory - short form. The UDI is a 6-question validated questionnaire assessing the urinary tract symptoms and their bothersomeness. Question three asks specifically about "Leakage related to activity, coughing, or sneezing", i.e. stress urinary incontinence. A low score indicates a minimal degree of severity impact
  units on a scale | 3 [2 to 3]
UDI score [Median (Inter-Quartile Range); unit: units on a scale] — Urogenital Distress inventory - short form. The UDI is a 6-question validated questionnaire assessing the urinary tract symptoms and their bothersomeness. Answers are scored from 0-3 (3 most bothersome). An average score is then obtained, ranging from 0-3.
  units on a scale | 1.5 [1.2 to 2]
MCS12 [Mean (Standard Deviation); unit: units on a scale] — The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. The questions were combined, scored, and weighted to create two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of 12 questions and range from 0-100, where a 0 score indicates the lowest and 100 the highest level of health measured by the scales.
  In MCS section, we are looking at Mental Health composite score.
  units on a scale | 47.9 (11.1)
PCS12 [Mean (Standard Deviation); unit: units on a scale] — The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. The questions were combined, scored, and weighted to create two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of 12 questions and range from 0-100, where a 0 score indicates the lowest and 100 the highest level of health measured by the scales
  In PCS section, we are looking at Physical Health composite score.
  units on a scale | 51.2 (8.3)
Peak flow rate (ml/sec) [Mean (Standard Deviation); unit: ml/sec] — Patients void on a commode equipped with a flowmeter which measure the volume voided and its flow rate.
  ml/sec | 22.9 (15.1)
Post void residual (ml) [Mean (Standard Deviation); unit: ml] — The Post void Residual is measured at the end of void during urodynamic studies by measuring, using the UDS catheter already in place, the residual urine volume in the bladder
  ml | 19.6 (21)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 50% or More Reduction in Number of Incontinence Episode Per Week
Description: number of women who experienced 50% or more reduction in number of incontinence episode per week on diary while using the incontinence ring, compared to baseline period.
Time Frame: baseline and 4 weeks
Population: All participants who were randomized and fitted with a ring are included in this intent to treat analysis. Patients for whom a ring could not be successfully fitted were considered failure (<50%) improvement)
Measure: Count of Participants; unit: Participants
Groups:
- Incontinence Ring: participants completed a 1-week diary during the last of 4 weeks of ring use. Women who did not wear the ring were considered failures (<50% improvement from baseline)
- Controls: participants completed a 1-week diary during the last of 4 weeks of the 'no treatment' week. Failure is determined as <50% improvement from baseline.
Arm/Group | Incontinence Ring | Controls
Number analyzed (Participants) | 24 | 24
Participants | 14 | 10

2. Secondary Outcome: Score on Question 3 of UDI 6
Description: Score (0-3) of response to question #3 (stress incontinence specific) of Urogenital Distress inventory - short form. The UDI is a 6-question validated questionnaire assessing the urinary tract symptoms and their bothersomeness. Question three asks specifically about "Leakage related to activity, coughing, or sneezing", i.e. stress urinary incontinence. Answer is scored from 0-3 (3 most bothersome).
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Incontinence Ring: Use of incontinence ring
- Controls: no treatment
Arm/Group | Incontinence Ring | Controls
Number analyzed (Participants) | 24 | 24
units on a scale | 1 [0 to 2] | 3 [2 to 3]

3. Secondary Outcome: UDI Overall Score
Description: Urogenital Distress inventory - short form. The UDI is a 6-question validated questionnaire assessing the urinary tract symptoms and their bothersomeness. Answers are scored from 0-3 (3 most bothersome). An average score is then obtained, ranging from 0-3.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Incontinence Ring: participants completed the UDI questionnaire at the end of 4 weeks of ring use.
- Controls: participants completed the UDI questionnaire at the end of 4 weeks of the 'no treatment' week.
Arm/Group | Incontinence Ring | Controls
Number analyzed (Participants) | 24 | 24
units on a scale | 0.7 [0.1 to 1.2] | 1.3 [1.1 to 1.7]

4. Secondary Outcome: Objective Cure Rate
Description: Number of Participants Without Urinary Stress Incontinence During Provocation testing during urodynamic studies (UDS). Provocations included valsalva and cough, first at 300 ml while lying then standing, followed, if no leakage was seen, to provocations at maximum cystometric capacity while standing.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Incontinence Ring: UDS done with ring in situ. UDS was performed while using the ring, towards the end of the 4-week ring use period.
- No Treatment: UDS done without ring. All patients had UDS done without the ring prior to entry into the study. This UDS was considered to reflect the 'no treatment' period, although technically it was done at baseline. A UDS during the 'no treatment' period would have been ideal, but this would have represented an additional UDS testing that likely would not have differed from the baseline testing. All patients needed to have UDS-proven urodynamic stress incontinence as inclusion criteria.
Arm/Group | Incontinence Ring | No Treatment
Number analyzed (Participants) | 24 | 26
Participants | 0 | 0

5. Secondary Outcome: Urodynamic Effect of the Incontinence Ring on Flow Rate
Description: Peak flow rate (ml/sec) during uninstrumented uroflow. The 'no treatment' flow rate was obtained during baseline urodynamic studies (UDS) and the 'incontinence ring' flow rate was obtained at the end of the ring period for each participants, while wearing the ring.
Time Frame: baseline and at 4 weeks of ring use.
Measure: Mean (Standard Deviation); unit: ml/sec
Groups:
- Incontinence Ring: UDS done with ring in place
- no Treatment: All participants underwent UDS at baseline , when not wearing a ring. The flow rate obtained during this part of hte study is considered the 'no treatment' flow rate, irrespective of study arm.
Arm/Group | Incontinence Ring | no Treatment
Number analyzed (Participants) | 24 | 26
ml/sec | 24.1 (11.6) | 22.9 (15.1)

6. Secondary Outcome: Impact on I-QOL
Description: The I-QOL (Incontinence-Quality of Life) is a valid and reproducible self-administered measure for assessing quality of life of patients with urinary incontinence. Items are scored on a 4-point Likert response scale (very much, moderately, a little, not at all). Scoring the I-QOL questionnaire involves summing the responses into a single score. The sum score is transformed to a 0-100 scale, with a higher number representing a better quality of life
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Incontinence Ring Users: Use of incontinence ring
  incontinence ring (Milex): Incontinence ring fitted to patient's anatomy (by choosing appropriate size). It is worn continually for the duration of the treatment period.
  Intravaginal incontinence ring placed proximally in the posterior vaginal fornix. Knob located at mid-urethra.
- Controls: no intervention
Arm/Group | Incontinence Ring Users | Controls
Number analyzed (Participants) | 24 | 24
units on a scale | 89.1 [72.3 to 95.5] | 70.9 [56.4 to 84.5]

7. Secondary Outcome: Patient Acceptability (10 cm VAS)
Description: participants completed a 10 cm visual analogue scale at the end of 4 weeks of ring use, rating their pelvic discomfort on a 10 cm scale; 0= none, 10= max.
Time Frame: 4 weeks
Population: Women did not fill out this VAS when not wearing the incontinence ring.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Incontinence Ring: While wearing the incontinence ring,w omen were asked to fill out the VAS
Arm/Group | Incontinence Ring
Number analyzed (Participants) | 24
cm | 0.6 (0.9)

8. Secondary Outcome: Post Void Residual
Description: Post void residual measured by catheter after free flow uroflowmetry
Time Frame: The UDS while wearing the ring was done 2-4 weeks into the 'ring' treatment period, at patient's convenience, the UDS done at baseline was considered representative of "no treatment" UDS.
Population: All uroflow were obtained on arrival of the patient in the UDS suite and prior to instrumentation. patients were asked to arrive with a full bladder, but some did not, explaining the lower number of women with available results.
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Incontinence Ring Users: PVR done at UDS during uroflow while using ring
- no Treatment: PVR done at baseline UDS after uroflow. UDS was needed to determine baseline eligibility. We felt that this baseline UDS was representative of the "no treatment' UDS and therefore considered as such. Doing a third UDs during the "no treatment" period per se was deemed unnecessary and subjected patient to redundant testing.
Arm/Group | Incontinence Ring Users | no Treatment
Number analyzed (Participants) | 23 | 21
ml | 15.9 (19.1) | 51.5 (67.9)

ADVERSE EVENTS:
Time Frame: 10 weeks
Groups:
- Incontinence Ring: Use of incontinence ring
  incontinence ring (Milex): Incontinence ring fitted to patient's anatomy (by choosing appropriate size). It is worn continually for the duration of the treatment period.
  Intravaginal incontinence ring placed proximally in the posterior vaginal fornix. Knob located at mid-urethra.
- No Treatment: no intervention
Arm/Group | Incontinence Ring | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

LIMITATIONS AND CAVEATS:
small sample size. slow recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No